CLINICAL TRIAL: NCT05722210
Title: Prevalence and Development of Liver Dysfunction in Hematopoietic Stem Cell Transplant: A Prospective Natural History Study
Brief Title: Prevalence and Development of Liver Dysfunction in Hematopoietic Stem Cell Transplant
Status: Not yet recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000545; 000545-DK
Record Dates: First submitted 2023-02-09; First posted 2023-02-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09-16

CONDITIONS: Hematopoietic Stem Cell Transplant
Keywords: Liver Disease; Liver Dysfunction; Natural History
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults >= 18 years of age: undergoing evaluation for hematopoietic stem cell transplant at the NIH Clinical Center
- Children 3-17 years of age: undergoing evaluation for hematopoietic stem cell transplant at the NIH Clinical Center

SUMMARY:
Background:

Hematopoietic stem cell transplant (HSCT) is a common treatment for many cancers and other illnesses. But many people who have HSCT go on to develop liver dysfunction. Researchers want to know more about how and why this happens. In this natural history study, they will try to learn what factors lead to liver dysfunction; how underlying liver disease may affect the results of HSCT; and how HSCT may contribute to liver dysfunction.

Objective:

To understand the links between HSCT and liver dysfunction.

Eligibility:

Adults aged 18 years or older and children 3 to 17 years who are being evaluated for HSCT.

Design:

This study involves 11 visits in 4 years. Most visits will be in the first year.

Before and after their HSCT, participants will undergo these tests:

Physical exam, including blood tests and a test of heart function. Participants will provide stool samples.

Liver biopsies. Samples of liver tissue will be removed. This may be done either by inserting a needle through the right side of the chest, or with a thin tube threaded to the liver from a vein in the neck. Adult participants will undergo this procedure 2 times: once before the HSCT and once about a year later.

Imaging scans. Participants will lie on a bed that moves into either a cylinder or a donut-shaped machine.

Ultrasound. Participants will lie still. A probe that uses sound waves will be slid over their skin to get pictures of the liver.

Fibroscan exam. This is like an ultrasound that uses a special probe to measure the toughness of the liver.

...

DETAILED DESCRIPTION:
Study Description:

Liver dysfunction is common in patients that have undergone hematopoietic stem cell transplant (HSCT) and is associated with increased mortality. We aim to study the natural history of liver dysfunction in HSCT, what factors contribute to the development of liver dysfunction, and how underlying liver disease affects complications and outcomes of HSCT. We hypothesize that those patients with underlying liver disease or those who develop liver disease have increased morbidity and mortality compared to those without liver disease.

Objectives:

Primary Objective:

To determine whether, at 3 months (Visit 7) after transplant, patients with liver disease at transplant are more likely to have died or have a total bilirubin >=4 mg/dL than those without liver disease at transplant.

Secondary Objectives:

To understand the impact of liver disease in HSCT on morbidity/mortality.

To understand the development and progression of liver disease in hematopoietic stem cell transplant

Tertiary Objectives:

To identify predictive/protective factors associated with presence or absence of liver disease, and severity of liver disease in patients receiving hematopoietic stem cell transplant.

Endpoints:

Primary Endpoints:

* Death or total bilirubin >=4 mg/dL at 3 months (Visit 7) after the transplant
* Mortality rate

Secondary Endpoints:

* Morbidity/cause of death
* Development of portal hypertension and sequelae (i.e., ascites, variceal bleed, thrombocytopenia, elevated portal pressure)
* Development of liver failure (i.e., coagulopathy with an International Normalized Ration (INR) 1.5, and any degree of mental alteration (encephalopathy in a subject without preexisting cirrhosis and with an illness of < 26 weeks duration, including subjects with Wilson s disease, vertically acquired HBV, or autoimmune hepatitis per AASLD guidelines 2011)
* Rate of infection (type bacterial, viral fungal, location: central line, organ infection, sepsis, etc.)

Liver dysfunction, characterized by development of the following conditions:

* Synthetic dysfunction: Total bilirubin > 4 mg/dL (20-40% in HSCT recipients or INR > 1.5
* Portal hypertension: Presence/absence of any of the following will qualify as portal hypertension- ascites, collateral vessels, elevated portal pressure
* Liver injury: ALT>4 times the upper limit of normal (22 IU/L in women, 29 IU/L in men) or Alkaline phosphatase >2.5 times the upper limit of normal

Tertiary Endpoints:

* Imaging, laboratory analysis of liver dysfunction, liver tissue pathology, medications/treatment course will be reviewed.
* Tertiary studies include stool microbiome studies, metabolomics, microbial translocation markers, flow cytometry, transcriptomics, growth factor measurement, cytokines, and chemokines measurement.

ELIGIBILITY:
* INCLUSION CRITERIA:

An individual who meets any of the following criteria will be included in this study:

* Male and female adults >=18 years of age and children 3-17 years of age
* Undergoing evaluation for hematopoietic stem cell transplant at the NIH Clinical Center

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this

study:

* Pregnancy or lactation
* Unable to comply with study procedures
* Inability to provide written informed consent

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: male and female subjects: adults 18 years of age and older, children 3-17 years of age undergoing hematopoietic stem cell transplant at the National Institutes of Health.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Death or total bilirubin >=4 at 91 days after the transplant | 91 days after transplant
  To determine whether, at 91 days after transplant, patients with liver disease at transplant are more likely to have died or have a total bilirubin >=4 than those without liver disease at transplant.
Mortality rate | 91 days after transplant
  To determine whether, at 91 days after transplant, patients with liver disease at transplant are more likely to have died or have a total bilirubin >=4 than those without liver disease at transplant.

SECONDARY OUTCOMES:
Rate of infection (type: bacterial, viral, fungal; location: central line, organ infection, sepsis, etc.) | 91 days after transplant
Development of portal hypertension and sequelae (i.e., ascites, variceal bleed, thrombocytopenia, elevated portal pressure) | 91 days after transplant
Morbitity/cause of death | 91 days after transplant
Development of liver failure | 91 days after transplant
  i.e., coagulopathy with an International Normalized Ratio (INR) 1.5, and any degree of mental alteration (encephalopathy) in a subject without preexisting cirrhosis and with an illness of <26 weeks duration, including patients with Wilson s disease, vertically acquired HBV, or autoimmune hepatitis per AASLD guidelines 2011.

CONTACTS AND LOCATIONS:
Overall Officials: Theo Heller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000545-DK.html